CLINICAL TRIAL: NCT04021199
Title: Screening for Genetic Forms of Diabetes in Convention of Care for Children and Adolescents With Diabetes (GENEPEDIAB)
Acronym: GENEPEDIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GENEPEDIAB
Record Dates: First submitted 2019-07-02; First posted 2019-07-16 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus; MODY
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1D Group (Active Comparator): * Retrospective analysis of data from active and historical diabetic patients within diabetes care conventions of pediatric endocrinology services; screening of patients with atypical diabetes; use of tests used in clinical routine to allow referral to the genetic diagnosis of the condition.
  * Prospective analysis of the evolution of new diabetic patients followed in pediatric endocrinology services of diabetes care conventions; screening of patients with atypical diabetes; use of tests used in clinical routine to allow the genetic diagnosis of the condition.
  * Screening of patients with atypical diabetes: first evaluated according to the "MODY" probability calculator. In addition, other clinical criteria will be used to improve the sensitivity and specificity of pediatric monogenic diabetes screening.
  Interventions: Genetic: Mody test
- MODY Group (Experimental): * Retrospective analysis of data from active and historical diabetic patients within diabetes care conventions of pediatric endocrinology services; screening of patients with atypical diabetes; use of tests used in clinical routine to allow referral to the genetic diagnosis of the condition.
  * Prospective analysis of the evolution of new diabetic patients followed in pediatric endocrinology services of diabetes care conventions; screening of patients with atypical diabetes; use of tests used in clinical routine to allow the genetic diagnosis of the condition.
  * Screening of patients with atypical diabetes: first evaluated according to the "MODY" probability calculator. In addition, other clinical criteria will be used to improve the sensitivity and specificity of pediatric monogenic diabetes screening.
  Interventions: Genetic: Mody test

INTERVENTIONS:
Genetic: Mody test — Subjects will be screened using a MODY gene-sequencing test, which includes GCK, HNF1A, HNF4A, HNF1B, KCNJ11, ABCC8, and INS gene sequencing.
  More comprehensive genetic tests will be conducted in patients without anomalies found after the MODY gene-sequencing test.

SUMMARY:
Background/Aims: Diabetes, which affects 420 million people worldwide with a continuously rising incidence, is defined by a state of chronic hyperglycemia; a criterion referring to a heterogeneous group of diseases with various etiologies and distinct therapeutic options. Besides the two main forms of diabetes (i.e., type 1 (T1D) and type 2 (T2D)), there are rare subtypes of the disease called monogenic diabetes (or formerly MODY) that are hardly diagnosed because of their resemblance to T1D or T2D. Since these monogenic diabetes may appear early in life, a consortium of expert pediatric clinical centers was created under a clinical research initiative (the GENEPEDIAB study) to develop tools for accurate diagnosis of rare diabetes and to propose appropriate care to these children and adolescents wrongly assigned to T1D or T2D cohorts. The GENEPEDIAB study was initiated in the context of a broader collaborative project (DiaType) with the objective to develop personalized diabetes medicine and better patient care.

Methods: For discrimination of patients with monogenic diabetes from those with classical forms of diabetes using the MODY probability calculator, patients enrolled in the GENEPEDIAB study are phenotyped and genotyped for T1D risk (anti-islet antibodies and HLA). Patients fulfilling sufficient criteria are then genotyped using the routine MODY panel, before being proposed a thorough gene analysis. More comprehensive genetic tests will be conducted in patients without anomalies found after the MODY gene-sequencing test.

Perspective: the GENEPEDIAB study will enable the investigators to adapt treatment to diabetes etiology and help to provide genetic counseling to patients and their family members. The investigators anticipate that its broad genetic analyses will provide them with important information about the genetic susceptibility of these subgroups of patients with atypical diabetes.

DETAILED DESCRIPTION:
BACKGROUND:

Diabetes currently affects 420 million people worldwide, a number that is expected to increase to 642 million in 2040. This disease is responsible for a high morbidity rate and an overall mortality equivalent to 5 million deaths per year. In Belgium, the prevalence of diabetes is estimated at 8% in adults over 35 years of age, the risk of diabetes being 3 to 5 times higher in populations with high consanguinity, mainly due to the susceptibility to generate recessive genetic variants, which are characteristic of atypical forms of diabetes.

Although diabetes is linearly defined by a state of chronic hyperglycaemia, this criterion refers to a heterogeneous group of diseases of various aetiologies and distinct therapeutic options. Ten to 15% of diabetic patients have insulin-dependent type 1 diabetes (T1D), attributed to autoimmune destruction of insulin-producing beta cells, while 80% of patients have type 2 diabetes (T2DM), treated - inter alia - with oral antidiabetic drugs. Despite the diagnosis of T1D is confirmed by the determination of specific antibodies, DT1 and T2D are clinically characterized by the phenotypic type and evolution of the patient, without recourse to specific etiological and/or pathognomonic criteria. Recently, subtypes of T1D and T2D have been categorized to help the clinician choose the best therapeutic interventions for the patient (i.e., dietary approach, physical activity, oral antidiabetic drugs, insulin, combined therapies).

Monogenic causes of diabetes are less common (up to 5% of all cases) and of recent discovery, their molecular basis having been established in the 1990s, under the name "maturity onset diabetes of the young" (MODY). The diagnosis of a genetic origin of diabetes has multiple consequences, primarily at therapeutic level. Despite the implications of a monogenic diabetes diagnosis, this form remains largely underdiagnosed, and it is accepted that 2 to 3% of active patients within diabetes conventions of care suffer from undetected genetic forms.

AIM:

Screening, using routinely diagnostic tools, of monogenic forms of diabetes in cohorts of paediatric patients with atypical forms of diabetes, who are followed in conventions of care for diabetic patients. After diagnosis of monogenic forms of diabetes, screened patients will be monitored and treated according to international recommendations applied to specifically recognized forms of diabetes.

The aim of GENEPEDIAB study is to improve the diagnosis of atypical forms of diabetes in children and adolescents, and not to evaluate the effects of treatment modification following genetic screening.

INTERVENTION:

1. Retrospective analysis of data from active and historical diabetic patients within diabetes care conventions of paediatric endocrinology services; screening of patients with atypical diabetes; use of clinical routine tests to allow genetic diagnosis of the condition.
2. Prospective analysis of the evolution of new diabetic patients followed in paediatric diabetes care conventions; screening of patients with atypical diabetes; use of clinical routine tests to allow genetic diagnosis of the condition.
3. Screening of patients with atypical diabetes:

   * The monogenic diabetes probability will initially be assessed using the MODY probability calculator (old terminology for monogenic diabetes), which identifies at risk patients based on clinical history (age, sex, body mass index, HbA1C, type of therapy, presence of diabetes in the family). This calculator is available on Internet at www.diabetesgenes.org.
   * In addition, other clinical criteria will be used to improve the sensitivity and specificity of screening for monogenic diabetes.
4. Genetic diagnosis of the condition:

   * The diagnosis of T1D will first be completed based on factors currently recognized by the International Society for Paediatric and Adolescent Diabetes (ISPAD): anti islet antibodies and at risk HLA genotype. Residual insulin secretion will be also evaluated.
   * Subjects that are detected using criteria described above will be screened using the routine MODY gene sequencing test, which includes GCK, HNF1A, HNF4A, HNF1B, KCNJ11, ABCC8, and INS gene sequencing.
   * More comprehensive genetic tests will be conducted in patients without anomalies found after the MODY gene-sequencing test.

PARTICIPATING SITES:

GENEPEDIAB is a multicentre study that include various diabetes care conventions of paediatric endocrinology services in Belgium.

* Main site: Cliniques universitaires Saint-Luc (UCLouvain), Brussel (Belgium)

  * Principal investigator : Dr. Philippe Lysy, Paediatric Endocrinology Unit
  * Co-investigators : PhD student Sophie Welsch, PhD Caroline Daems, Paediatric Endocrinology Unit
  * Clinical Research Coordinator : Paola Gallo, Paediatric Endocrinology Unit
* Other sites:

  * CHU ND-des Bruyeres (ULg), Liege (Belgium) - Prof. Marie-Christine Lebrethon;
  * CHU UCL Namur site Mont-Godinne & CHU UCL Namur site Sainte-Elisabeth (UCLouvain), Namur (Belgium) - Dr. Dominique Beckers & Dr. Thierry Mouraux;
  * CHC, Liege (Belgium) - Dr. Nicole Seret;
  * Grand Hopital de Charleroi site Notre Dame (GHdC), Charleroi (Belgium) - Dr. Jacques Louis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 18 years at the age of diabetes diagnosis.
* Patients followed and/or diagnosed within diabetes care agreements of the pediatric endocrinology departments participating in the study.

Exclusion Criteria:

* none

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 446 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Diagnostic of atypical diabetes using follow-up of clinical parameters: Weight | At diabetes diagnosis
  Weight in kilograms (Kg)
Diagnostic of atypical diabetes using follow-up of clinical parameters: Height | At diabetes diagnosis
  Height in meters (m)
Diagnostic of atypical diabetes using follow-up of clinical parameters: BMI | At diabetes diagnosis
  Body Mass Index (Kg/m²)
Diagnostic of atypical diabetes using follow-up of laboratory results: HbA1c (%) | from diabetes diagnosis to study inclusion. (The study inclusion will be from 18 months after diagnosis to several years)
  Glicated hemoglobin (%)
Diagnostic of atypical diabetes using follow-up of laboratory results: HbA1c (mmol/mol) | from diabetes diagnosis to study inclusion. (The study inclusion will be from 18 months after diagnosis to several years)
  Glicated hemoglobin (mmol/mol)
Diagnostic of atypical diabetes using follow-up of laboratory results: Glycaemia | from diabetes diagnosis to study inclusion
  Glycaemia (mg/dL)
Diagnostic of atypical diabetes using follow-up of laboratory results: C-peptide | from diabetes diagnosis to study inclusion. (The study inclusion will be from 18 months after diagnosis to several years)
  C-peptide (pmol/mL)
Genetic diagnosis of diabetes: Anti-islets antibodies | from diabetes diagnosis to study inclusion. (The study inclusion will be from 18 months after diagnosis to several years)
  Presence of measurable Anti-islets antibodies
Genetic diagnosis of diabetes: HLA genotype | from diabetes diagnosis to study inclusion. (The study inclusion will be from 18 months after diagnosis to several years)
  Presence of at risk HLA genotype
Genetic diagnosis of atypical diabetes: MODY gene-sequencing test | at inclusion in the study
  MODY gene-sequencing test (GCK, HNF1A, HNF4A, HNF1B, KCNJ11, ABCC8, and INS gene sequencing)
Genetic diagnosis of atypical diabetes: More comprehensive genetic tests | After MODY gene-sequencing test, from 3 months to 1.5 year after study inclusion
  More comprehensive genetic tests will be conducted in patients without anomalies found after the MODY gene-sequencing test.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lysy, Principal Investigator — Cliniques universitaires Saint-Luc - UCLouvain
Locations (1):
- Cliniques universitaires Saint-Luc - UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No